CLINICAL TRIAL: NCT04619147
Title: Invasive Fungal Infections in Patients Following Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: QA/64470/PMCC-2020
Record Dates: First submitted 2020-10-04; First posted 2020-11-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Invasive Fungal Infections; Stem Cell Transplant Complications
Keywords: Posaconazole; Antifungal prophylaxis; Invasive fungal infections; Epidemiology; Allogeneic haematopoiectic stem cell transplant
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without invasive fungal infections (IFI): This will be our control cohort. Most of the patients would have been on posaconazole prophylaxis.
  Interventions: Other: No intervention
- Patients with invasive fungal infections (IFI): This will be the group that we will be interested in. IFI would be diagnosed based on EORTC/ MSG definitions, and most of them would have been on posaconazole prophylaxis. Underlying risk factors of acquiring IFI in this cohort of patients will be compared with that of the control cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is descriptive, retrospective study to evaluate the epidemiology of invasive fungal infections (IFI) in patients undergoing allogeneic haematopoiectic stem cell transplant in the era of antifungal prophylaxis with posaconazole delay-released tablets.

SUMMARY:
This study will be a descriptive, retrospective evaluation and analysis of invasive fungal infections (IFI) conducted in patients who underwent allogeneic haematopoiectic stem cell transplant (aHSCT) in a single tertiary transplant centre, the Bone Marrow Transplant Clinical Service across Peter MacCallum Cancer Centre (PMCC) and Royal Melbourne Hospital (RMH), Victoria, Australia.

DETAILED DESCRIPTION:
Invasive fungal infections (IFIs) remain a leading cause of mortality and morbidity in immunosuppressed patients who undergo allogenic haematopoiectic stem cell transplant (aHSCT). Both yeast and moulds cause serious IFIs in this cohort of patients, especially during the pre-engraftment neutropenic phase, and post-engraftment period when patients need to be on prolonged course of corticosteroids for severe graft-versus-host-disease (GVHD). Other risk factors for IFIs include environmental factors, genetic factors, and co-viral infections. Candida spp accounts for most of the invasive yeast infections whereas Aspergillus spp is the most common mould in aHSCT recipients. The estimated incidence of proven and probable invasive Candida infections without antifungal prophylaxis ranged from 8% to 24%; on the other hand the incidence of invasive aspergillosis was reported to be in between 3% to 14%. IFIs are often associated with mortality rate as high as 60%, and have been identified as one of the independent predictors of death in multivariate analysis. Other complications include extended hospital stay from invasive fungal infections, intensive care admissions, huge treatment cost and significant morbidity and reduced quality of life in patients.

Antifungal prophylaxis with fluconazole in aHSCT recipient has become a routine in the 1990s after several studies demonstrated fits efficacy in reducing morbidity and mortality in this group of patients. In 2007 two multi-centres, double-blinded trials, involving either aHSCT patients with GVHD or non-transplantation patients with haematologic malignancy and prolonged neutropenia, proved superiority of the mould-active agent with posaconazole to fluconazole in preventing invasive aspergillosis and death from IFI. This finding was further confirmed by a systemic review and meta-analysis in 2012 that included 20 randomised trials, comparing mould-active prophylaxis with fluconazole prophylaxis in aHSCT recipients or patients with haematologic malignancy receiving chemotherapy. Consequently, current Australian guideline proposed that all patients at high risk of IFIs (>10%) be administered mould-active antifungal prophylaxis, and these patients include aHSCT recipients with expected neutropenia of >14 days, extensive chronic GVHD, severe steroid refractory or dependent GVHD and patients with acute leukaemia or myelodysplasia who are undergoing induction or re-induction chemotherapy. Broad-spectrum triazole posaconazole is the recommended first-line therapy, with other triazoles such as voriconazole, itraconazole or echinocandin as alternative therapy.

In Australia, until 2015 posaconazole was only available in liquid form. Posaconazole suspension needs to be taken with high-fat meal or supplements to enhance its absorption. The unpredictable absorption of the suspension, especially in patients with mucositis or neutropenic colitis from chemotherapy prompted the recommendation of monitoring the trough posaconazole level. However in Victoria, this assay was not widely available and the turnaround time was often long, hence it could not be performed in real-time fashion for optimal management. A delayed-release tablet formulation of posaconazole was approved by TGA in 2013 and it was added to the Pharmaceutical Benefits Scheme (PBS) in Australia in mid-2015. At the same time an intravenous formulation was also approved by TGA. The tablet formulation has improved bioavailability as its absorption was not dependent upon high fat or supplement content like its liquid counterpart, and it is anticipated that its administration will likely result in therapeutic drug levels. As a result routine therapeutic drug monitoring is not required during prophylaxis with posaconazole tablets. The availability of the intravenous and tablet formulation may have a positive impact on the rates of IFIs, however this has not been formally reviewed in Australia. Patients on posaconazole prophylaxis with the Bone Marrow Transplant Clinical Service are currently on either tablets or the intravenous formulation (if patients have factors that impaired oral intake).

Although the introduction of mould-active antifungal prophylaxis has reduced the incidence of IFIs significantly, there have been numerous studies reporting on the changing epidemiology of these infections and concerns raised over the rates of breakthrough IFIs and emergence of azole-resistant strains, including non-albicans species of invasive candidiasis. Winston et al reported of a breakthrough IFI rate 7.5% while on posaconazole liquid formulation, and this finding was consistent with some European studies, which found incidence of 3-14% of breakthrough invasive mould disease. On the other hand, Tverdek et al reported a much improved rate of breakthrough IFI of 2% in 343 patients who received intravenous or delay-released tablet formulation of posaconazole, suggesting that these new formulations resulted in better absorption of the medication with direct implication on rates of IFI.

Most of the studies mentioned above, that reported incidence of IFIs in the era of mold-active antifungal prophylaxis, were conducted in the United States or Europe. Specifically there has not been a study done locally in Australia looking at this question, including breakthrough IFIs. The epidemiology of fungal isolates in Australia may be very different compared to that of European or American continents. For example there have been reports of higher incidence of systemic infection due to Lomentospora prolificans in Australia and Spain, involving patients with acute leukemia or with aHSCT.

The introduction of the posaconazole tablets may have improved IFI breakthrough rates in our local Bone Marrow Transplant Centre, although this has not yet been examined. Anecdotal evidence suggests that the rates of posaconazole therapeutic drug monitoring at our institution are low, but again this has not been formally documented.

It is imperative to evaluate the epidemiology of these infections in this cohort in the new era of posaconazole prophylaxis, to monitor the rates of breakthrough IFIs and if there is emergence of azole-resistance fungal isolates in the Australian context. This study aims to establish an overview of IFIs in patients receiving stem cell transplant. Not only will it provide invaluable information on local epidemiology and microbiology of invasive fungal infections, it will also enable more appropriate planning of antifungal prophylaxis strategies in these high-risk patients.

Study's hypothesis:

* Invasive fungal infections remain an ongoing challenge and one of leading sources of morbidity and mortality post allogeneic haematopoietic stem cell transplant (aHSCT) despite the widespread use of anti-mould prophylaxis.
* Improvements could be made in the prophylaxis, treatment and monitoring of fungal infections.
* Knowledge of local epidemiology could inform efforts to improve current practice.

Aims of the study:

1. To describe the epidemiology of invasive fungal infections (IFIs) in patients undergoing allogeneic haematopoiectic stem cell transplant (aHSCT) in the era of antifungal prophylaxis with posaconazole delay-released tablets.
2. To report the incidence of IFIs, and in particular breakthrough IFIs in this cohort of high-risk patients.
3. To identify the risk factors of acquiring IFIs in this cohort of patients.
4. To evaluate the current practice and use of antifungal agents as prophylaxis, the reasons for selection, the frequency of therapeutic drug monitoring, adverse effects and appropriateness of antifungal prescription.
5. To determine the all-cause mortality rate and fungal infections related death following aHSCT at 3, 6 and 12 months post aHSCT.
6. To identify areas of current divergence from best practice in the prevention and treatment of invasive fungal infections in patients receiving allogeneic HCT.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are above 18 years of age,
* Who underwent allogeneic haematopoietic stem cell transplant (aHSCT) from 1 January 2017 to 1 January 2019 with the Bone Marrow Transplant Clinical Service at Royal Melbourne Hospital (RMH) & Peter MacCallum Cancer Centre (PMCC), Victoria, Australia
* Only the first transplant procedure will be included in the analysis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent allogeneic haematopoiectic stem cell transplant (aHSCT) in a single tertiary transplant centre, the Bone Marrow Transplant Clinical Service across Peter MacCallum Cancer Centre (PMCC) and Royal Melbourne Hospital (RMH), Victoria, Australia.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Incidence of invasive fungal infections (IFI) in patients | One year
  Incidence of IFI will be calculated as number of new episodes of IFI (index episode only) during the data collection period (1 Jan 2017 to 1 Jan 2019) over total number of patients who have undergone allogeneic stem cell transplant during the same period.

SECONDARY OUTCOMES:
Breakthrough rates of invasive fungal infections (IFI) | one year
  Breakthrough IFI is defined as any IFI occurring during exposure to an antifungal drug, including fungi outside the spectrum of activity of an antifungal. Incidence of breakthrough rates of IFI will be calculated as number of episodes IFI over number of courses of anti fungal prophylaxis in a defined period.
Mortality | One year
  To determine all-cause mortality, non-relapse mortality and infection-related mortality in this cohort of patients.
Current practice of antifungal prophylaxis | one year
  Number of patients on different types of antifungal prophylaxis during a defined period. For patients who were on antifungal prophylaxis which required therapeutic drug monitoring (TDM)- proportion of patients who actually had TDM done and proportion of patients whose TDM was within therapeutic level.
Adverse effects from antifungal prescription | One year
  Number of participants with adverse events from antifungal as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
De-identified demographics data of patients, transplant characteristic, details of invasive fungal infections

REFERENCES:
- [Background] Wingard JR. The changing face of invasive fungal infections in hematopoietic cell transplant recipients. Curr Opin Oncol. 2005 Mar;17(2):89-92. doi: 10.1097/01.cco.0000152975.65477.7c. PMID 15725910
- [Background] Wingard JR, Hsu J, Hiemenz JW. Hematopoietic stem cell transplantation: an overview of infection risks and epidemiology. Infect Dis Clin North Am. 2010 Jun;24(2):257-72. doi: 10.1016/j.idc.2010.01.010. PMID 20466269
- [Background] Grow WB, Moreb JS, Roque D, Manion K, Leather H, Reddy V, Khan SA, Finiewicz KJ, Nguyen H, Clancy CJ, Mehta PS, Wingard JR. Late onset of invasive aspergillus infection in bone marrow transplant patients at a university hospital. Bone Marrow Transplant. 2002 Jan;29(1):15-9. doi: 10.1038/sj.bmt.1703332. PMID 11840139
- [Background] Yong MK, Ananda-Rajah M, Cameron PU, Morrissey CO, Spencer A, Ritchie D, Cheng AC, Lewin SR, Slavin M. Cytomegalovirus Reactivation Is Associated with Increased Risk of Late-Onset Invasive Fungal Disease after Allogeneic Hematopoietic Stem Cell Transplantation: A Multicenter Study in the Current Era of Viral Load Monitoring. Biol Blood Marrow Transplant. 2017 Nov;23(11):1961-1967. doi: 10.1016/j.bbmt.2017.07.025. Epub 2017 Aug 7. PMID 28797778
- [Background] Girmenia C, Raiola AM, Piciocchi A, Algarotti A, Stanzani M, Cudillo L, Pecoraro C, Guidi S, Iori AP, Montante B, Chiusolo P, Lanino E, Carella AM, Zucchetti E, Bruno B, Irrera G, Patriarca F, Baronciani D, Musso M, Prete A, Risitano AM, Russo D, Mordini N, Pastore D, Vacca A, Onida F, Falcioni S, Pisapia G, Milone G, Vallisa D, Olivieri A, Bonini A, Castagnola E, Sica S, Majolino I, Bosi A, Busca A, Arcese W, Bandini G, Bacigalupo A, Rambaldi A, Locasciulli A. Incidence and outcome of invasive fungal diseases after allogeneic stem cell transplantation: a prospective study of the Gruppo Italiano Trapianto Midollo Osseo (GITMO). Biol Blood Marrow Transplant. 2014 Jun;20(6):872-80. doi: 10.1016/j.bbmt.2014.03.004. Epub 2014 Mar 14. PMID 24631738
- [Background] Cornely OA, Gachot B, Akan H, Bassetti M, Uzun O, Kibbler C, Marchetti O, de Burghgraeve P, Ramadan S, Pylkkanen L, Ameye L, Paesmans M, Donnelly JP; EORTC Infectious Diseases Group. Epidemiology and outcome of fungemia in a cancer Cohort of the Infectious Diseases Group (IDG) of the European Organization for Research and Treatment of Cancer (EORTC 65031). Clin Infect Dis. 2015 Aug 1;61(3):324-31. doi: 10.1093/cid/civ293. Epub 2015 Apr 13. PMID 25870323
- [Background] Marr KA, Carter RA, Boeckh M, Martin P, Corey L. Invasive aspergillosis in allogeneic stem cell transplant recipients: changes in epidemiology and risk factors. Blood. 2002 Dec 15;100(13):4358-66. doi: 10.1182/blood-2002-05-1496. Epub 2002 Aug 22. PMID 12393425
- [Background] Marr KA, Carter RA, Crippa F, Wald A, Corey L. Epidemiology and outcome of mould infections in hematopoietic stem cell transplant recipients. Clin Infect Dis. 2002 Apr 1;34(7):909-17. doi: 10.1086/339202. Epub 2002 Feb 26. PMID 11880955
- [Background] Rotstein C, Bow EJ, Laverdiere M, Ioannou S, Carr D, Moghaddam N. Randomized placebo-controlled trial of fluconazole prophylaxis for neutropenic cancer patients: benefit based on purpose and intensity of cytotoxic therapy. The Canadian Fluconazole Prophylaxis Study Group. Clin Infect Dis. 1999 Feb;28(2):331-40. doi: 10.1086/515128. PMID 10064252
- [Background] Wald A, Leisenring W, van Burik JA, Bowden RA. Epidemiology of Aspergillus infections in a large cohort of patients undergoing bone marrow transplantation. J Infect Dis. 1997 Jun;175(6):1459-66. doi: 10.1086/516480. PMID 9180187
- [Background] Ceesay MM, Sadique Z, Harris R, Ehrlich A, Adams EJ, Pagliuca A. Prospective evaluation of the cost of diagnosis and treatment of invasive fungal disease in a cohort of adult haematology patients in the UK. J Antimicrob Chemother. 2015 Apr;70(4):1175-81. doi: 10.1093/jac/dku506. Epub 2014 Dec 21. PMID 25535218
- [Background] Ananda-Rajah MR, Cheng A, Morrissey CO, Spelman T, Dooley M, Neville AM, Slavin M. Attributable hospital cost and antifungal treatment of invasive fungal diseases in high-risk hematology patients: an economic modeling approach. Antimicrob Agents Chemother. 2011 May;55(5):1953-60. doi: 10.1128/AAC.01423-10. Epub 2011 Feb 28. PMID 21357302
- [Background] Goodman JL, Winston DJ, Greenfield RA, Chandrasekar PH, Fox B, Kaizer H, Shadduck RK, Shea TC, Stiff P, Friedman DJ, et al. A controlled trial of fluconazole to prevent fungal infections in patients undergoing bone marrow transplantation. N Engl J Med. 1992 Mar 26;326(13):845-51. doi: 10.1056/NEJM199203263261301. PMID 1542320
- [Background] Slavin MA, Osborne B, Adams R, Levenstein MJ, Schoch HG, Feldman AR, Meyers JD, Bowden RA. Efficacy and safety of fluconazole prophylaxis for fungal infections after marrow transplantation--a prospective, randomized, double-blind study. J Infect Dis. 1995 Jun;171(6):1545-52. doi: 10.1093/infdis/171.6.1545. PMID 7769290
- [Background] Dykewicz CA; National Center for Infectious Diseases, Centers for Disease Control and Prevention; Infectious Diseases Society of America; American Society for Blood and Marrow Transplantation. Guidelines for preventing opportunistic infections among hematopoietic stem cell transplant recipients: focus on community respiratory virus infections. Biol Blood Marrow Transplant. 2001;7 Suppl:19S-22S. doi: 10.1053/bbmt.2001.v7.pm11777100.
- [Background] Ullmann AJ, Lipton JH, Vesole DH, Chandrasekar P, Langston A, Tarantolo SR, Greinix H, Morais de Azevedo W, Reddy V, Boparai N, Pedicone L, Patino H, Durrant S. Posaconazole or fluconazole for prophylaxis in severe graft-versus-host disease. N Engl J Med. 2007 Jan 25;356(4):335-47. doi: 10.1056/NEJMoa061098. PMID 17251530
- [Background] Cornely OA, Maertens J, Winston DJ, Perfect J, Ullmann AJ, Walsh TJ, Helfgott D, Holowiecki J, Stockelberg D, Goh YT, Petrini M, Hardalo C, Suresh R, Angulo-Gonzalez D. Posaconazole vs. fluconazole or itraconazole prophylaxis in patients with neutropenia. N Engl J Med. 2007 Jan 25;356(4):348-59. doi: 10.1056/NEJMoa061094. PMID 17251531
- [Background] Ethier MC, Science M, Beyene J, Briel M, Lehrnbecher T, Sung L. Mould-active compared with fluconazole prophylaxis to prevent invasive fungal diseases in cancer patients receiving chemotherapy or haematopoietic stem-cell transplantation: a systematic review and meta-analysis of randomised controlled trials. Br J Cancer. 2012 May 8;106(10):1626-37. doi: 10.1038/bjc.2012.147. PMID 22568999
- [Background] Ananda-Rajah MR, Grigg A, Slavin MA. Making sense of posaconazole therapeutic drug monitoring: a practical approach. Curr Opin Infect Dis. 2012 Dec;25(6):605-11. doi: 10.1097/QCO.0b013e328359a56e. PMID 23086185
- [Background] Fleming S, Yannakou CK, Haeusler GM, Clark J, Grigg A, Heath CH, Bajel A, van Hal SJ, Chen SC, Milliken ST, Morrissey CO, Tam CS, Szer J, Weinkove R, Slavin MA. Consensus guidelines for antifungal prophylaxis in haematological malignancy and haemopoietic stem cell transplantation, 2014. Intern Med J. 2014 Dec;44(12b):1283-97. doi: 10.1111/imj.12595. PMID 25482741
- [Background] Dekkers BGJ, Bakker M, van der Elst KCM, Sturkenboom MGG, Veringa A, Span LFR, Alffenaar JC. Therapeutic Drug Monitoring of Posaconazole: an Update. Curr Fungal Infect Rep. 2016;10:51-61. doi: 10.1007/s12281-016-0255-4. Epub 2016 May 7. PMID 27358662
- [Background] van Hal SJ, Gilroy NM, Morrissey CO, Worth LJ, Szer J, Tam CS, Chen SC, Thursky KA, Slavin MA. Survey of antifungal prophylaxis and fungal diagnostic tests employed in malignant haematology and haemopoietic stem cell transplantation (HSCT) in Australia and New Zealand. Intern Med J. 2014 Dec;44(12b):1277-82. doi: 10.1111/imj.12594. PMID 25482740
- [Background] Cornely OA, Duarte RF, Haider S, Chandrasekar P, Helfgott D, Jimenez JL, Candoni A, Raad I, Laverdiere M, Langston A, Kartsonis N, Van Iersel M, Connelly N, Waskin H. Phase 3 pharmacokinetics and safety study of a posaconazole tablet formulation in patients at risk for invasive fungal disease. J Antimicrob Chemother. 2016 Mar;71(3):718-26. doi: 10.1093/jac/dkv380. Epub 2015 Nov 26. PMID 26612870
- [Background] Winston DJ, Bartoni K, Territo MC, Schiller GJ. Efficacy, safety, and breakthrough infections associated with standard long-term posaconazole antifungal prophylaxis in allogeneic stem cell transplantation recipients. Biol Blood Marrow Transplant. 2011 Apr;17(4):507-15. doi: 10.1016/j.bbmt.2010.04.017. Epub 2010 May 9. PMID 20460163
- [Background] Auberger J, Lass-Florl C, Aigner M, Clausen J, Gastl G, Nachbaur D. Invasive fungal breakthrough infections, fungal colonization and emergence of resistant strains in high-risk patients receiving antifungal prophylaxis with posaconazole: real-life data from a single-centre institutional retrospective observational study. J Antimicrob Chemother. 2012 Sep;67(9):2268-73. doi: 10.1093/jac/dks189. Epub 2012 May 30. PMID 22653819
- [Background] Lerolle N, Raffoux E, Socie G, Touratier S, Sauvageon H, Porcher R, Bretagne S, Bergeron A, Azoulay E, Molina JM, Lafaurie M. Breakthrough invasive fungal disease in patients receiving posaconazole primary prophylaxis: a 4-year study. Clin Microbiol Infect. 2014 Nov;20(11):O952-9. doi: 10.1111/1469-0691.12688. Epub 2014 Jul 12. PMID 24861577
- [Background] Lamoth F, Chung SJ, Damonti L, Alexander BD. Changing Epidemiology of Invasive Mold Infections in Patients Receiving Azole Prophylaxis. Clin Infect Dis. 2017 Jun 1;64(11):1619-1621. doi: 10.1093/cid/cix130. PMID 28199491
- [Background] Kimura M, Araoka H, Yamamoto H, Asano-Mori Y, Nakamura S, Yamagoe S, Ohno H, Miyazaki Y, Abe M, Yuasa M, Kaji D, Kageyama K, Nishida A, Ishiwata K, Takagi S, Yamamoto G, Uchida N, Izutsu K, Wake A, Taniguchi S, Yoneyama A. Clinical and Microbiological Characteristics of Breakthrough Candidemia in Allogeneic Hematopoietic Stem Cell Transplant Recipients in a Japanese Hospital. Antimicrob Agents Chemother. 2017 Mar 24;61(4):e01791-16. doi: 10.1128/AAC.01791-16. Print 2017 Apr. PMID 28115352
- [Background] Tverdek FP, Heo ST, Aitken SL, Granwehr B, Kontoyiannis DP. Real-Life Assessment of the Safety and Effectiveness of the New Tablet and Intravenous Formulations of Posaconazole in the Prophylaxis of Invasive Fungal Infections via Analysis of 343 Courses. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00188-17. doi: 10.1128/AAC.00188-17. Print 2017 Aug. PMID 28507111
- [Background] Wood GM, McCormack JG, Muir DB, Ellis DH, Ridley MF, Pritchard R, Harrison M. Clinical features of human infection with Scedosporium inflatum. Clin Infect Dis. 1992 May;14(5):1027-33. doi: 10.1093/clinids/14.5.1027. PMID 1534693